CLINICAL TRIAL: NCT04936321
Title: Enhancing the Efficacy of Migraine Self-Management in Children with Comorbid Insomnia
Brief Title: Intervention for Sleep and Pain in Youth: a Randomized Controlled Trial
Acronym: I-SPY-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Principal Investigator, Emily Law, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00003090
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Insomnia; Migraine Disorders; Headache Disorders
Keywords: pediatric; children; adolescent; sleep; pain; headache; cognitive-behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Migraine Disorders; Headache Disorders; Pain; Headache | interventions — Pain Management

STUDY DESIGN:
Intervention Model Description: The study design is a two arm, two-phase RCT. In Phase 1, the effects of internet-delivered CBT insomnia intervention will be compared to internet-delivered sleep education control. In Phase 2, all participants will receive internet-delivered CBT pain intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Because all study procedures delivered online, neither study participants nor investigators. care providers, or outcomes assessors will have knowledge of the treatment assignment and thus this trial can be carried out as a double-blinded RCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Education + CBT for Pain (Active Comparator): Participants will receive access to internet-delivered sleep education during Phase 1 (6 weeks) of the study followed by internet-delivered CBT for pain management during Phase 2 (6 weeks) of the study.
  Interventions: Behavioral: Internet-delivered CBT for Pain Management; Behavioral: Internet-delivered Sleep Education
- CBT for Insomnia + CBT for Pain (Experimental): Participants will receive access to internet-delivered CBT for insomnia during Phase 1 (6 weeks) of the study followed by internet-delivered CBT for pain management during Phase 2 (6 weeks) of the study.
  Interventions: Behavioral: Internet-delivered CBT for Insomnia; Behavioral: Internet-delivered CBT for Pain Management

INTERVENTIONS:
Behavioral: Internet-delivered CBT for Insomnia — The program delivers the core components of CBT for insomnia including sleep hygiene, stimulus control, and sleep restriction. Treatment duration is 6 weeks.
  Arms: CBT for Insomnia + CBT for Pain
Behavioral: Internet-delivered CBT for Pain Management — The program delivers the core components of CBT for pain management including: pain education, training in behavioral and cognitive pain coping skills, instruction in increasing activity participation, and training in parental operant and communication strategies. Treatment duration is 6 weeks.
  Other Names: Web-MAP (Web-based Management of Adolescent Pain)
Behavioral: Internet-delivered Sleep Education — The program delivers publicly available information about sleep.
  Arms: Sleep Education + CBT for Pain

SUMMARY:
Insomnia is a common comorbidity among adolescents with migraine. This randomized controlled clinical trial aims to determine efficacy of cognitive-behavioral therapy (CBT) for insomnia, as well as the combined effect of CBT insomnia and pain interventions, on reducing insomnia symptoms and headache-related disability in adolescents with migraine. The long-term goal is to offer effective, tailored self-management interventions that can address migraine and co-morbid sleep problems in adolescence and disrupt a cycle of persistent, disabling migraine from continuing into adulthood.

DETAILED DESCRIPTION:
This aims of this study are to: 1) test efficacy of cognitive-behavioral therapy (CBT) insomnia intervention for youth with migraine and comorbid insomnia, and 2) investigate how changes in sleep may modify response to CBT pain intervention. Participants will include 250 youth and their parents. Youth will be ages 11-17 years, with migraine (with or without aura, chronic migraine) and comorbid insomnia. In Phase 1, participants will be randomly assigned to receive access to internet-delivered CBT insomnia intervention or internet-delivered sleep education control over 6 weeks. In Phase 2, all participants will receive access to internet-delivered CBT pain intervention over 6 weeks. Assessments will occur at baseline, immediately after Phase 1 intervention, immediately after Phase 2 intervention, and 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old
* Headache present for at least three months and insomnia symptoms for the past month
* Access to the Internet on any web-enabled device

Exclusion Criteria:

* Non-English speaking
* Diagnosed sleep disorder (e.g. sleep apnea, narcolepsy)
* Unable to read at 5th grade level or complete surveys independently
* A serious comorbid chronic condition (e.g., diabetes, arthritis, cancer)

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia symptoms | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The 7-item Insomnia Severity Index (ISI) measures severity of insomnia symptoms. Total scores above 8 on the ISI indicate clinically significant insomnia in adult and adolescent samples.
Change in headache-related disability | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The CALI-9 is a 9-item self-report instrument of headache-related disability in children and adolescents that measures difficulty in performing usual daily physical, social, and recreational activities. The measure will be completed daily for 14 days at baseline, after phase 1, after phase 2, and 6-month follow-up

SECONDARY OUTCOMES:
Change in sleep quality | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The Adolescent Sleep Wake Scale-Short Form (ASWS) is a 10-item measure. The total score indicates overall perception of sleep quality.
Change in sleep patterns | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  14-days of actigraphic monitoring with the Actiwatch Spectrum Plus to assess minutes of estimated sleep, wake time after sleep onset, and sleep efficiency.
Change in headache frequency | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The number of headache days reported each day for 14 days.
Change in headache pain intensity | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  11-point numerical rating scale with anchors of 0 = no pain to 10 = worst pain possible. Reported each day for 14 days.
Change in anxiety symptoms | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The Generalized Anxiety Disorder-7 is a 7-item measure. The total score indicates anxiety severity over the last two weeks.
Change in depressive symptoms | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The Patient Health Questionnaire-9 is a 9 item measure. The total score indicates severity of depression over the last two weeks.
Change in health-related quality of life as assessed by the Pediatric Quality of Life Inventory 4.0 | Baseline, immediately after treatment phase 1, immediately after treatment phase 2, 6-month follow-up
  The Pediatric Quality of Life Inventory 4.0. is a measure of health-related quality of life. The total score indicates perceived mental and physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Law, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Law EF, Ritterband L, Zhou C, Palermo TM. Intervention for Sleep and Pain in Youth (ISPY-RCT): protocol for a two-phase randomized controlled trial of sequenced cognitive-behavioral therapy for insomnia and pain management in adolescents with migraine. Trials. 2023 Jan 12;24(1):25. doi: 10.1186/s13063-022-07035-9. PMID 36635741